CLINICAL TRIAL: NCT02486224
Title: Metabolomic Analysis of the Impacts of Hydration Status on Exercise Performance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 shutdown prevented study enrollment. Staff was subsequently lost to execute trial aims.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1502689413
Record Dates: First submitted 2015-06-08; First posted 2015-07-01 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Dehydration; Physical Exertion; Salivary Osmolar Concentration; Urinary Osmolar Concentration
Keywords: deep sea mineral water; exercise recovery; hydration; salivary osmolar concentration; urinary osmolar concentration
MeSH Terms: conditions — Dehydration | interventions — gatorade

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Kona Deep (Experimental): Subjects will receive Kona Deep post-exercise
  Interventions: Dietary Supplement: Kona Deep
- Spring Water (Placebo Comparator): Subjects will receive commercially available Spring Water post-exercise
  Interventions: Dietary Supplement: Spring Water
- Sports Drink (Active Comparator): Subjects will receive commercially available Sports Drink post-exercise
  Interventions: Dietary Supplement: Sports Drink

INTERVENTIONS:
Dietary Supplement: Kona Deep — Subjects will receive Kona Deep post exercise
  Other Names: Deep Seawater
  Arms: Kona Deep
Dietary Supplement: Spring Water — Subjects will receive Spring Water post exercise
  Arms: Spring Water
Dietary Supplement: Sports Drink — Subjects will receive Sports Drink post exercise
  Other Names: Gatorade
  Arms: Sports Drink

SUMMARY:
Kona Deep is bottled water extracted from a depth of 3000 feet off the cost of Kona, Hawaii. Kona Deep claims that this unique source provides water that is "naturally free of pathogens, chemicals and pollutants and rich in nutrients and minerals that are readily absorbed by the body". The investigators wish to examine Kona Deep's claim that this water is "beneficial to the human body" by testing the impact of drinking Kona Deep on exercise performance and recovery. Subjects will be exercised to a safe level of dehydration and then will be rehydrated with Kona Deep water, or commercially available bottled spring water or Gatorade as controls. Subjects will perform a simple exercise to evaluate peak power performance. This measurement will be compared between rehydration methods for significant differences.

DETAILED DESCRIPTION:
Exercise-induced dehydration is very common in athletes and regularly active individuals. Hypohydration, if sufficiently severe, can negatively impact physical performance and mental capacity. Development of an efficient rehydration therapy could prove beneficial in these circumstances. Multiple animal studies have shown the positive effects of desalinated deep-sea mineral water on various physiological conditions. The beneficial effects of deep-sea mineral water may be attributed to its unique mineral composition, particularly magnesium, which is highly abundant in deep-sea water. The investigators wish to evaluate whether a similar response occurs in post-exercise rehydration using deep ocean water from a different source. Kona Deep is marketed as Hawaiian glacier water drawn from a depth of 915 m off the Kona coast that is naturally rich in electrolytes and nutrients, and that is free of mercury, harmful bacterial, and pollutants, making it a desired drinking water source. Accordingly, the investigators will investigate whether subjects administered Kona Deep following an exercise challenge undergo more rapid rehydration and demonstrate higher peak power production compared to subjects administered commercially available liquids. Euhydrated subjects in this study will be exposed to an exercise-challenge protocol (stationary biking) under warm conditions (30°C) to accelerate dehydration. Dehydration will be measured as a body mass loss of 3-5% (maximum exercise time will be 180 minutes). A body mass loss of 3% is the minimal amount lost during a similar exercise-dehydration protocol but where significance was still observed in exercise performance, recovery, and physiological parameters. During the post-exercise recovery period, subjects will consume one of three liquids in a volume equivalent to 1.5 times the body mass lost. Rehydration measured by salivary and urinary osmolality and exercise recovery will be measured such as oxygen consumption (VO2) at 60% estimated maximal heart rate and peak power production by contraction of the knee extensors before exercise, immediately after exercise, and after the rehydration period.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers, BMI: 18.5-24.9, 20-25 years of age, physically active

Exclusion Criteria:

* prescription medications, BMI > 24.9

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Osmolar Concentration during Exercise, Post-Exercise, Post-Rehydration | 0-180 minutes
  Saliva will be collected at regular intervals throughout the study protocol

SECONDARY OUTCOMES:
Change in Urinary Osmolar Concentration during Exercise, Post-Exercise, Post-Rehydration | 0-180 minutes
  Urine will be collected prior to, immediately following exercise and immediately following rehydration.
Change in Lower body muscle power Pre-Exercise, Post-Exercise, Post-Rehydration | 0-180 minutes
  Lower body muscle power will be determined prior to, immediately following exercise and immediately following rehydration. This will be executed using a Biodex Dynamometer to determine single leg extension and flexion torque.

CONTACTS AND LOCATIONS:
Overall Officials: John P Konhilas, PhD, Principal Investigator — University of Arizona
Locations (1):
- Ina A. Gittings Building, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The University of Arizona (UA) will assure the timely release and sharing of data no later than the acceptance for publication of the main findings from the final dataset and will protect the rights and privacy of human subjects who participate in NIH sponsored research by redacting all identifiers and adoption of other strategies to minimize risks of unauthorized disclosure of personal identifiers in accordance with authorization and consent documents. UA will share data resulting from sponsored projects with research colleagues by depositing data on a secure web-accessible data warehouses or arranging distribution of data, reagents, protein targets, and protocols to other researchers using established mechanisms and repositories. Manuscripts will be submitted for publication in high-quality peer-reviewed journals, adhering to NIH Public Access Policy guidelines. Additionally, findings will be presented and discussed at relevant national conferences.

REFERENCES:
- [Background] Miyamura M, Yoshioka S, Hamada A, Takuma D, Yokota J, Kusunose M, Kyotani S, Kawakita H, Odani K, Tsutsui Y, Nishioka Y. Difference between deep seawater and surface seawater in the preventive effect of atherosclerosis. Biol Pharm Bull. 2004 Nov;27(11):1784-7. doi: 10.1248/bpb.27.1784. PMID 15516723
- [Background] Tsuchiya Y, Watanabe A, Fujisawa N, Kaneko T, Ishizu T, Fujimoto T, Nakamura K, Yamamoto M. Effects of desalted deep seawater on hematologic and blood chemical values in mice. Tohoku J Exp Med. 2004 Jul;203(3):175-82. doi: 10.1620/tjem.203.175. PMID 15240926
- [Background] Katsuda S, Yasukawa T, Nakagawa K, Miyake M, Yamasaki M, Katahira K, Mohri M, Shimizu T, Hazama A. Deep-sea water improves cardiovascular hemodynamics in Kurosawa and Kusanagi-Hypercholesterolemic (KHC) rabbits. Biol Pharm Bull. 2008 Jan;31(1):38-44. doi: 10.1248/bpb.31.38. PMID 18175939
- [Background] Bohl CH, Volpe SL. Magnesium and exercise. Crit Rev Food Sci Nutr. 2002;42(6):533-63. doi: 10.1080/20024091054247. PMID 12487419
- [Background] Hou CW, Tsai YS, Jean WH, Chen CY, Ivy JL, Huang CY, Kuo CH. Deep ocean mineral water accelerates recovery from physical fatigue. J Int Soc Sports Nutr. 2013 Feb 12;10(1):7. doi: 10.1186/1550-2783-10-7. PMID 23402436
- [Background] Galloway SD, Maughan RJ. Effects of ambient temperature on the capacity to perform prolonged cycle exercise in man. Med Sci Sports Exerc. 1997 Sep;29(9):1240-9. doi: 10.1097/00005768-199709000-00018. PMID 9309637
- [Background] Munoz CX, McKenzie AL, Armstrong LE. Optimal hydration biomarkers: consideration of daily activities. Obes Facts. 2014;7 Suppl 2(Suppl 2):13-8. doi: 10.1159/000360655. Epub 2014 Apr 4. No abstract available. PMID 24853347
- [Derived] Harris PR, Keen DA, Constantopoulos E, Weninger SN, Hines E, Koppinger MP, Khalpey ZI, Konhilas JP. Fluid type influences acute hydration and muscle performance recovery in human subjects. J Int Soc Sports Nutr. 2019 Apr 4;16(1):15. doi: 10.1186/s12970-019-0282-y. PMID 30947727